CLINICAL TRIAL: NCT04971135
Title: A Phase 1 Study to Assess the Safety and Tolerability of Single and Multiple Ascending Doses of SAN711 in Healthy Participants
Brief Title: First-in-human Study of SAN711 in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saniona (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SAN711-01
Record Dates: First submitted 2021-07-02; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SAN711 (SAD) (Experimental): 6 out of 8 participants per cohort (up to 7 cohorts) will be randomized to receive a single dose of SAN711
  Interventions: Drug: SAN711
- Placebo (SAD) (Placebo Comparator): 2 out of 8 participants per cohort (up to 7 cohorts) will be randomized to receive a single dose of Placebo
  Interventions: Other: Placebo
- SAN711 (MAD) (Experimental): 6 out of 8 participants per cohort (up to 3 cohorts) will be randomized to receive 14 daily doses of SAN711
  Interventions: Drug: SAN711
- Placebo (MAD) (Placebo Comparator): 2 out of 8 participants per cohort (up to 3 cohorts) will be randomized to receive 14 daily doses of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SAN711 — SAN711 liquid formulation
  Arms: SAN711 (MAD); SAN711 (SAD)
Other: Placebo — Matching placebo
  Arms: Placebo (MAD); Placebo (SAD)

SUMMARY:
Phase 1, first-in-human, double-blind, randomized, placebo-controlled, parallel group, single ascending dose (SAD) and multiple ascending dose (MAD) study

ELIGIBILITY:
Inclusion Criteria:

* Healthy, determined by Screening medical evaluation (medical history, physical examination, vital signs, safety 12-lead electrocardiogram [ECG], and clinical laboratory evaluations, including liver and renal function tests which must be within normal limits)
* Body mass index (BMI) between 18.5 and 29.9 kg/m2, inclusive at Screening
* Non-smoker (and no other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (<500 ng/mL) at the Screening Visit and admission
* Female participants must be women of non-childbearing potential (WONCBP); defined as follows: surgically sterile (ie, had a hysterectomy, or bilateral oophorectomy, or bilateral salpingectomy ≥6 months prior to the first dose of study drug); or Postmenopausal (no menses) for at least 1 year prior to the first dose of study drug. Postmenopausal status must be confirmed by FSH testing at screening

Exclusion Criteria:

* Participant has a history or evidence of any clinically significant cardiovascular, general gastrointestinal, endocrine, hematologic, hepatic, immunological, metabolic, urologic, pulmonary, neurological, dermatologic, psychiatric, renal, and/or other major disease or malignancy as judged by the investigator
* Participant answers "yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the "Suicidal Behavior" portion of the Columbia Suicide Severity Rating Scale
* Participant's current alcohol intake exceeds 14 units/week for men and women (1 unit = half pint of beer, 1 glass of wine, 1 measure of spirits)
* Participant is unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to check-in Day and until final discharge Day inclusive
* Participant is unwilling to avoid consumption of caffeine-containing beverages within 48 hours prior to day of admission until final discharge day
* Participant has a history of illicit substance use OR a positive urine drug test (eg, cocaine, amphetamines, methylenedioxymethamphetamine (MDMA), barbiturates, opiates, benzodiazepines, or cannabinoids) or urine alcohol test at the Screening Visit or admission
* Participant has a positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C, or HBsAg negative/anti-HBc positive/anti-HBs negative, or human immunodeficiency virus (HIV) 1 and/or -2 antibodies
* At Screening and Baseline, systolic blood pressure (SBP) greater than 140 or less than 90 mm Hg, or diastolic blood pressure (DBP) greater than 90 or less than 40 mm Hg, in the supine position, at screening or baseline. Borderline values (ie values that are within 5 mm Hg for blood pressure or 5 beats/min for heart rate) will be repeated. Subjects can be included if the repeat value is within range or still borderline, but deemed not clinically significant by the investigator
* Corrected QT interval using Fridericia's formula >450 msec for males and >470 msec for females
* Resting bradycardia (heart rate [HR] <40 beats per minute [bpm]) or tachycardia (HR >100 bpm)
* Personal or family history of congenital long QT syndrome or sudden death
* Screening or Admission ECG with QRS and/or T wave judged to be unfavorable for a consistently accurate QT measurement (eg, neuromuscular artifact that cannot be readily eliminated, arrhythmias, indistinct QRS onset, low amplitude T wave, merged T- and U-waves, prominent U waves)
* Evidence of atrial fibrillation, atrial flutter, complete branch block, Wolf-Parkinson-White Syndrome, or cardiac pacemaker at screening or on admission
* Receipt of COVID-19 vaccine within 2 weeks prior to baseline or scheduled for vaccination during the study
* COVID-19 infection within 90 days of screening or evidence of current COVID-19 infection within the past 4 weeks at screening, between screening and admission, or at admission
* If unvaccinated for COVID-19, contact with an individual with COVID-19 infection in the past 14 days at screening, between screening and admission, or at admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events (TEAEs) [SAD] | Initiation of dosing through 96 hours post dosing
  Incidence of TEAEs during SAD
TEAEs [MAD] | Initiation of dosing through 16 days post dosing
  Incidence of TEAEs during MAD
Adverse Events of Special Interest (AESIs) [SAD] | Initiation of dosing through 96 hours post dosing
  Incidence of AESIs during SAD
AESIs [MAD] | Initiation of dosing through 16 days post dosing
  Incidence of AESIs during MAD

SECONDARY OUTCOMES:
PK Parameters: Cmax [SAD] | Baseline (Predose) through 96 hours post dosing
  Maximum observed plasma concentration at Tmax during SAD
PK Parameters: Cmax [MAD] | Day 1 (Predose) through Day 16
  Maximum observed plasma concentration at Tmax during MAD
PK Parameters: Tmax [SAD] | Baseline (Predose) through 96 hours post dosing
  Time of maximum observed plasma concentration during SAD
PK Parameters: Tmax [MAD] | Day 1 (Predose) through Day 16
  Time of maximum observed plasma concentration during MAD
PK Parameters: t1/2 [SAD] | Baseline (Predose) through 96 hours post dosing
  Apparent terminal phase half-life during SAD
PK Parameters: t1/2 [MAD] | Day 1 (Predose) through Day 16
  Apparent terminal phase half-life during MAD
PK Parameters: AUC-last [SAD] | Baseline (Predose) through 96 hours post dosing
  Area under the plasma concentration time curve from time zero to T-last, the time at which Last measurable plasma concentration (C-last) is observed during SAD
PK Parameters: AUC-last [MAD] | Day 1 (Predose) through Day 16
  Area under the plasma concentration time curve from time zero to T-last, the time at which Last measurable plasma concentration (C-last) is observed during MAD
PK Parameters: AUC-inf [SAD] | Baseline (Predose) through 96 hours post dosing
  Area under the plasma concentration time curve extrapolated to infinity during SAD
PK Parameters: AUC-inf [MAD] | Day 1 (Predose) through Day 16
  Area under the plasma concentration time curve extrapolated to infinity during MAD

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will consider requests for access to SAN711-01 Study materials following completion of SAN711 Development
Supporting Information: Study Protocol, SAP, ICF, CSR